CLINICAL TRIAL: NCT04785001
Title: Assessment of New Physiological, Radiological and Activity Markers in Patients Treated by Spinal Cord Stimulation for Chronic Lower Limb Pain
Brief Title: New Markers to Assess the Efficacity of Spinal Cord Stimulation for the Treatment of Chronic Lower Limb Pain (MOTIVE)
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: HBD_2020_23
Record Dates: First submitted 2021-01-26; First posted 2021-03-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Stimulation
Keywords: SCS (spinal cord stimulation); HRV (Heart Rate Variability); MRIf (anatomical and functional magnetic resonance imaging)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
By combining the usual care of patients eligible for spinal cord stimulation (SME) with measurements of the HRV index (Heart Rate Variability), objective measurements of activity (number of steps, quality of sleep) and measurements of connectivity obtained by anatomical and functional magnetic resonance imaging (fMRI), the collection of preliminary data necessary for the analysis of markers correlated with the efficiency of stimulation will be possible. Ultimately, these markers could be used to optimize the perioperative management of these patients.

DETAILED DESCRIPTION:
The rebellious chronic neuropathic pain of the lower limbs (including the sequelae lumbosciatica) causes a major functional repercussion and an impairment of the quality of life. Spinal cord stimulation (SCS) is offered when other treatments are ineffective or insufficient (K. Kumar et al., 2007). This technique has been used in routine care for over 20 years, with a well-established clinical benefit for these indications, and recognized by HAS (see 2014 recommendations in appendix 1). Moreover, recent technical progress has made it possible to provide better user comfort for implanted patients, in particular with new stimulation methods that best adapt to the activities and feelings of the patients (De Ridder & Vanneste, 2016; V . Kumar et al., 2018).

The therapeutic objectives defined between the candidate patient for EMS and the Pain team are part of a personalized rehabilitation and reintegration process. This is to reduce the pain felt by the patient but also the functional impact, by gradually resuming activity, taking into account the specific situation of each patient. Functional limitation depends on several factors, such as exercise deconditioning but also fear of movement that is essential to assess in patients who are candidates for EMS. Patient care involves an assessment made by a trained multi-professional team in which the role of the pain coordinator (IDEC) is central, with therapeutic education work through regular physical and telephone consultations. Self-administered questionnaires analyzing functional abilities, quality of life and pain are currently being used for the pre- and post-operative assessment of patients undergoing EMS. Although they are a diagnostic and decision-making tool, they nevertheless correspond to a subjective assessment of the patient of his abilities as he sees them, and not to an assessment of his actual objective abilities. Thus, despite the technical progress represented by the new stimulation methods, the perioperative assessment of patients treated for EMS lacks personalized tools.

The recent development of technological tools that are easy to use on a daily basis, such as activity trackers and smartwatches, is an attractive option in chronic pathologies, but still insufficiently used in current medical practice. A review of the literature has shown the value of the use of activity trackers, particularly in postoperative follow-up and functional rehabilitation (Appelboom et al., 2016), and in low back pain patients (GORDON & BLOXHAM, 2017 ). Another study evaluating the data collected by an actimeter integrated into a stimulation generator compared to the patient's verbal report on his activities reports an overestimation of the functional impact by patients in self-evaluation (Goudman et al., 2018). Likewise, a study on the evaluation of the quality of sleep highlighted a difference between the feelings reported by the patient, the self-questionnaires and the data recorded in polysomnography (Jaeger et al., 2019), with a trend to increase sleep disorders. All of these studies confirm the limits in terms of the reliability of declarative data and the need for objective measures to assess the symptoms of patients in chronic conditions.

In addition, some of these devices have recently made it possible to evaluate the vmHRV (vagally-mediated Heart Rate Variability) index (Hernando et al., 2018). This physiological index has been studied for MOTIVE_Protocole_v1_20200610 HBD_2020_23 IDRCB 2020-A01731-38 11/40 several years, and has shown its interest in various chronic pathologies such as depression, cardiovascular pathologies, fibromyalgia (Kemp et al., 2010). Thus, compared to healthy control subjects, patients with chronic pain have a decreased vmHRV index linked to lower vagal activity (Koenig et al., 2016). In addition, in chronic pain patients, a correlation was observed between taking analgesics, the impact of pain on daily life and a significantly reduced vmHRV index. Moreover, patients with little relief from drug treatment had the lowest vmHRV index (Koenig et al., 2015), thus showing a link between this index and the severity of chronic pain, its daily impact, l effectiveness of drug treatment. Likewise, a correlation has been demonstrated between the degree of catastrophization of pain in patients and the vmHRV index (Koenig et al., 2016). Finally, a recent review of the imaging data associated with the measurement of the HRV index suggests a link between functional connectivity and the activity of certain brain regions (ventral striatum, anterior cingulate cortex, medial pre-frontal cortex, putamen ), the ability to manage stress and emotions, and the HRV index (Thayer et al., 2012), thus proposing a neurovisceral integration model. The vmHRV index can therefore be considered as an objective marker in the assessment of emotional and physiological coping skills in a patient with chronic pain. This aspect is crucial in the evaluation and management of these patients, and more particularly when an invasive therapy is envisaged such as EMS.

Finally, the development of certain imaging sequences makes it possible to study the anatomical (diffusion tensor sequences: DTI) and functional (functional MRI sequences) connectivity in regions of interest in patients, in particular at rest (Fox & Raichle, 2007). During nociceptive stimulation, the functional activation of certain regions of interest was demonstrated, grouped together under the term "pain matrix": insula, primary and secondary somatosensory cortex, thalamus, anterior cingulate cortex, pre- frontal, tonsil and peri-acqueductal gray matter (Apkarian et al., 2005; Leknes & Tracey, 2008). Chronic pain alters the functioning of neural circuits in these regions, leading to changes in connectivity and activity observable in neuroimaging (Baliki et al., 2012; Wood et al., 2007). A prospective study conducted in 39 patients has also shown the predictive character of some of these changes during the chronicization of pain in a cohort of patients suffering from subacute low back pain (Baliki et al., 2012): patients developing pain patients (which lasts beyond 6 months) immediately presented an alteration in the functioning of the neural circuits involved in motivation, with a stronger anatomical and functional connectivity between the nucleus accumbens and the medial pre-frontal cortex, compared to the patients recovering from the subacute episode. Since then, other studies have suggested a link between the process of pain chronicization and changes in the anatomical and functional connectivity of cortico-striated circuits involved in cognitive and motivational aspects (Navratilova & Porreca, 2014). Activation of the meso-limbic motivational and reward circuit has also been shown to be involved in the perception of pain relief (Leknes et al., 2011; Navratilova et al., 2012; Seymour et al., 2005) .

The interest of these new cardiac markers (HRV), radiological (anatomical and functional connectivity in MRI) and activity (connected watch) in the management of patients eligible for stimulation medullary will be evaluate. The use of a connected watch continuously measuring activity (number of steps, distance covered), sleep (duration of deep and light sleep, number of nocturnal awakenings), and the HRV index could provide an objective assessment and complementary to the self-questionnaires and the usual interviews. The MRI profile of anatomical and functional connectivity in the regions of interest linked to chronic pain and motivation in patients treated for EMS, would allow to seek a link between functional outcome, motivation and the ability to adapt and manage stress.

By combining the usual care of patients eligible for an EMS with measurements of the HRV index, objective measurements of activity (number of steps, quality of sleep), and connectivity measurements obtained on MRI, the collection of preliminary data to identify markers correlated with the effectiveness of EMS will be possible. Ultimately, these markers could be used to optimize the perioperative management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb pain included in the inclusion criteria for spinal cord stimulation according to HAS recommendations: neuropathic, lumbar radicular sequelae after spinal surgery, complex regional pain syndrome (CRPS)
* Chronic pain that has been present for at least 6 months
* Rebellious pain resistant to drug and non-drug treatments well conducted;
* Functional impact defined by a score> 20% on the Oswestry scale;
* Patient affiliated or beneficiary of a social security scheme;
* Patient who consented to participate in the study.

Exclusion Criteria:

* Presence of a surgical contraindication to the implantation of material (chronic infection, long-term anticoagulant treatment that cannot be interrupted, contraindication to anesthesia);
* Addiction (according to DSM IV);
* Major depressive syndrome despite appropriate treatment and / or psychotic symptoms (according to DSM IV);
* Unbalanced psychiatric disorder;
* Intermittent pain or present for less than 6 months;
* Diffuse painful syndrome;
* Progressive disease, associated inflammatory rheumatic pathology, and any other disabling pathology limiting physical activity (advanced articular osteoarthritis);
* Absolute contraindication to MRI (e.g. pace-maker, implantable stimulator, intra-orbital metallic foreign body);
* Language barrier or cognitive disorders preventing understanding of the research protocol;
* Person benefiting from a legal protection measure;
* Pregnant or breastfeeding woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for drug-resistant neuropathic pain in the lower limbs and requiring implantation for SCS according to HAS criteria will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of Heart Rate Variability (HRV) in chronic lower leg pain patients treated with spinal cord stimulation. | 3 months after implantation
  Heart rate variability will be evaluated before (baseline) and 3 months after surgery. HRV parameters, including time domain and frequency domain, will be obtained from 24-hour Holter monitoring. Two time-domain variables will be used to determine HRV : the standard deviation of intervals of all normal beat (SDNN) and the root mean square of the difference of successive R-R intervals (rMSSD).

CONTACTS AND LOCATIONS:
Overall Officials: Hayat BELAID, Dr, Principal Investigator — Fondation Ophtalmologie Adolphe Rothschild
Locations (1):
- Fondation Ophtalmologie Adolphe de Rothschild, Paris, paris, France